CLINICAL TRIAL: NCT05546619
Title: Research on Effectiveness and Safety of the Treatment, Hyperthermic Intraperitoneal Chemotherapy Combined With Tislelizumab and Targeted Therapy, That is Used for High-risk Hepatocellular Carcinoma After R0 Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sulai Liu (Other)
Responsible Party: Sponsor-Investigator, Sulai Liu, Dc., Hunan Provincial People's Hospital
Organization: Hunan Provincial People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLiu
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: High-risk hepatocellular carcinoma; Adjuvant therapy; HIPEC; Tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treating with a Design Protocol (Experimental)
  Interventions: Drug: HIPEC+tislelizumab + targeted therapy

INTERVENTIONS:
Drug: HIPEC+tislelizumab + targeted therapy — Patients with open liver lobe/segment resection, tumor excision, lymph node dissection will receive medication.

SUMMARY:
There are limited treatment options for HCC with high recurrence risk, and there is no consistent plan for adjuvant therapy after surgery. Hence an unmet clinical need. Based on previous studies on unresectable HCC patients combined with targeted and immunotherapy, it has been found that the effect is significant, but the effect of combined with HIPEC is not clear, and no similar studies have been reported. Therefore, this project intends to carry out a single-arm clinical study on the efficacy and safety of HIPEC + tislelizumab combined with targeted therapy for high recurrence risk HCC. And observe the clinical benefits, to provide new ideas and evidence-based basis for the treatment of HCC with high recurrence risk.

ELIGIBILITY:
Inclusion Criteria:

* (1) In line with the diagnostic criteria of Western medicine, the pathological section was diagnosed as HCC; imaging and intraoperative exploration of HCC patients with high risk of recurrence: multiple tumors or satellite lesions, tumor diameter>5cm, HCC rupture and bleeding, combined with vascular invasion, and serum AFP>32ng/ml.

(2)18-70 years (3) Liver function: Child-Pugh A、B (4) Patients voluntarily receive treatment with this program.

Exclusion Criteria:

* (1) Patients did not meet the inclusion criteria. (2) Use of other antineoplastic drugs during the follow-up period (3) Severe heart and kidney damage. (4) Failure to follow the prescription for medication, and unable to judge the efficacy or incomplete information (5) Not suitable for targeted therapy and anti-PD1 immunotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
RFS | 1 year
  Relapse free survival

SECONDARY OUTCOMES:
OS | 10 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial People's Hospital(The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gentile D, Donadon M, Lleo A, Aghemo A, Roncalli M, di Tommaso L, Torzilli G. Surgical Treatment of Hepatocholangiocarcinoma: A Systematic Review. Liver Cancer. 2020 Jan;9(1):15-27. doi: 10.1159/000503719. Epub 2019 Nov 1. PMID 32071906
- [Result] Foerster F, Gairing SJ, Muller L, Galle PR. NAFLD-driven HCC: Safety and efficacy of current and emerging treatment options. J Hepatol. 2022 Feb;76(2):446-457. doi: 10.1016/j.jhep.2021.09.007. Epub 2021 Sep 20. PMID 34555422
- [Result] Satriano L, Lewinska M, Rodrigues PM, Banales JM, Andersen JB. Metabolic rearrangements in primary liver cancers: cause and consequences. Nat Rev Gastroenterol Hepatol. 2019 Dec;16(12):748-766. doi: 10.1038/s41575-019-0217-8. Epub 2019 Oct 30. PMID 31666728
- [Result] Ding X, He M, Chan AWH, Song QX, Sze SC, Chen H, Man MKH, Man K, Chan SL, Lai PBS, Wang X, Wong N. Genomic and Epigenomic Features of Primary and Recurrent Hepatocellular Carcinomas. Gastroenterology. 2020 May 16:S0016-5085(20)30659-4. doi: 10.1053/j.gastro.2019.09.056. Online ahead of print. PMID 32428506
- [Result] Li X, Ramadori P, Pfister D, Seehawer M, Zender L, Heikenwalder M. The immunological and metabolic landscape in primary and metastatic liver cancer. Nat Rev Cancer. 2021 Sep;21(9):541-557. doi: 10.1038/s41568-021-00383-9. Epub 2021 Jul 29. PMID 34326518
- [Result] Wang H, Lu Z, Zhao X. Tumorigenesis, diagnosis, and therapeutic potential of exosomes in liver cancer. J Hematol Oncol. 2019 Dec 9;12(1):133. doi: 10.1186/s13045-019-0806-6. PMID 31815633
- [Result] Sharma SA, Kowgier M, Hansen BE, Brouwer WP, Maan R, Wong D, Shah H, Khalili K, Yim C, Heathcote EJ, Janssen HLA, Sherman M, Hirschfield GM, Feld JJ. Toronto HCC risk index: A validated scoring system to predict 10-year risk of HCC in patients with cirrhosis. J Hepatol. 2017 Aug 24:S0168-8278(17)32248-1. doi: 10.1016/j.jhep.2017.07.033. Online ahead of print. PMID 28844936
- [Result] Bhatt A, de Hingh I, Van Der Speeten K, Hubner M, Deraco M, Bakrin N, Villeneuve L, Kusamura S, Glehen O. HIPEC Methodology and Regimens: The Need for an Expert Consensus. Ann Surg Oncol. 2021 Dec;28(13):9098-9113. doi: 10.1245/s10434-021-10193-w. Epub 2021 Jun 17. PMID 34142293
- [Result] Pameijer CR. HIPEC Trials and the US: A Review and Call to Action. Ann Surg Oncol. 2022 Feb;29(2):866-872. doi: 10.1245/s10434-021-10769-6. Epub 2021 Oct 1. No abstract available. PMID 34599434
- [Result] Blumenthaler AN, Allen CJ, Ikoma N, Blum M, Das P, Minsky BD, Mansfield PF, Ajani JA, Badgwell BD. Laparoscopic HIPEC for Low-Volume Peritoneal Metastasis in Gastric and Gastroesophageal Adenocarcinoma. Ann Surg Oncol. 2020 Dec;27(13):5047-5056. doi: 10.1245/s10434-020-08968-8. Epub 2020 Jul 31. PMID 32737700
- [Result] Klempner SJ, Ryan DP. HIPEC for colorectal peritoneal metastases. Lancet Oncol. 2021 Feb;22(2):162-164. doi: 10.1016/S1470-2045(20)30693-8. Epub 2021 Jan 18. No abstract available. PMID 33476594
- [Result] van Stein RM, Aalbers AGJ, Sonke GS, van Driel WJ. Hyperthermic Intraperitoneal Chemotherapy for Ovarian and Colorectal Cancer: A Review. JAMA Oncol. 2021 Aug 1;7(8):1231-1238. doi: 10.1001/jamaoncol.2021.0580. PMID 33956063
- [Result] Strijker D, Meijerink WJHJ, Bremers AJA, de Reuver P, van Laarhoven CJHM, van den Heuvel B. Prehabilitation to improve postoperative outcomes in patients with peritoneal carcinomatosis undergoing hyperthermic intraperitoneal chemotherapy (HIPEC): A scoping review. Eur J Surg Oncol. 2022 Mar;48(3):657-665. doi: 10.1016/j.ejso.2021.10.006. Epub 2021 Oct 20. PMID 34702591
- [Result] Gulmez S, Polat E, Duman U, Senger AS, Uzun O, Ozduman O, Oz A, Subasi IE, Duman M. Hepatic bridge and round ligament of the liver during cytoreductive surgery: a retrospective cohort. Langenbecks Arch Surg. 2022 May;407(3):1201-1207. doi: 10.1007/s00423-021-02386-4. Epub 2021 Nov 29. PMID 34845541
- [Result] Liu S, Zhong Z, Yi W, Yu Z, Zhang Z, Xia G, Jiang B, Song Y, Peng C. Effect of Hyperthermic Intraperitoneal Perfusion Chemotherapy Combined with Radical Surgery and Capecitabine on Stage III Gallbladder Cancer. Can J Gastroenterol Hepatol. 2021 Oct 8;2021:4006786. doi: 10.1155/2021/4006786. eCollection 2021. PMID 34660468
- [Result] Riley RS, June CH, Langer R, Mitchell MJ. Delivery technologies for cancer immunotherapy. Nat Rev Drug Discov. 2019 Mar;18(3):175-196. doi: 10.1038/s41573-018-0006-z. PMID 30622344
- [Result] O'Donnell JS, Teng MWL, Smyth MJ. Cancer immunoediting and resistance to T cell-based immunotherapy. Nat Rev Clin Oncol. 2019 Mar;16(3):151-167. doi: 10.1038/s41571-018-0142-8. PMID 30523282
- [Result] Marabelle A, Tselikas L, de Baere T, Houot R. Intratumoral immunotherapy: using the tumor as the remedy. Ann Oncol. 2017 Dec 1;28(suppl_12):xii33-xii43. doi: 10.1093/annonc/mdx683. PMID 29253115
- [Result] Ziogas IA, Evangeliou AP, Giannis D, Hayat MH, Mylonas KS, Tohme S, Geller DA, Elias N, Goyal L, Tsoulfas G. The Role of Immunotherapy in Hepatocellular Carcinoma: A Systematic Review and Pooled Analysis of 2,402 Patients. Oncologist. 2021 Jun;26(6):e1036-e1049. doi: 10.1002/onco.13638. Epub 2021 Jan 2. PMID 33314549
- [Result] Osarogiagbon RU. Tislelizumab-A Promising New Option for Enhancing Chemotherapy Benefit in Treatment for Advanced Squamous Cell Lung Cancer. JAMA Oncol. 2021 May 1;7(5):717-719. doi: 10.1001/jamaoncol.2021.0262. No abstract available. PMID 33792622
- [Result] Lee A, Keam SJ. Tislelizumab: First Approval. Drugs. 2020 Apr;80(6):617-624. doi: 10.1007/s40265-020-01286-z. PMID 32185681
- [Result] Yi M, Zheng X, Niu M, Zhu S, Ge H, Wu K. Combination strategies with PD-1/PD-L1 blockade: current advances and future directions. Mol Cancer. 2022 Jan 21;21(1):28. doi: 10.1186/s12943-021-01489-2. PMID 35062949
- [Result] Shen L, Guo J, Zhang Q, Pan H, Yuan Y, Bai Y, Liu T, Zhou Q, Zhao J, Shu Y, Huang X, Wang S, Wang J, Zhou A, Ye D, Sun T, Gao Y, Yang S, Wang Z, Li J, Wu YL. Tislelizumab in Chinese patients with advanced solid tumors: an open-label, non-comparative, phase 1/2 study. J Immunother Cancer. 2020 Jun;8(1):e000437. doi: 10.1136/jitc-2019-000437. PMID 32561638
- [Result] Kissel M, Berndt S, Fiebig L, Kling S, Ji Q, Gu Q, Lang T, Hafner FT, Teufel M, Zopf D. Antitumor effects of regorafenib and sorafenib in preclinical models of hepatocellular carcinoma. Oncotarget. 2017 Nov 6;8(63):107096-107108. doi: 10.18632/oncotarget.22334. eCollection 2017 Dec 5. PMID 29291014
- [Result] Saraswati S, Alhaider A, Abdelgadir AM, Tanwer P, Korashy HM. Phloretin attenuates STAT-3 activity and overcomes sorafenib resistance targeting SHP-1-mediated inhibition of STAT3 and Akt/VEGFR2 pathway in hepatocellular carcinoma. Cell Commun Signal. 2019 Oct 16;17(1):127. doi: 10.1186/s12964-019-0430-7. PMID 31619257
- [Result] Matsuki M, Hoshi T, Yamamoto Y, Ikemori-Kawada M, Minoshima Y, Funahashi Y, Matsui J. Lenvatinib inhibits angiogenesis and tumor fibroblast growth factor signaling pathways in human hepatocellular carcinoma models. Cancer Med. 2018 Jun;7(6):2641-2653. doi: 10.1002/cam4.1517. Epub 2018 May 7. PMID 29733511
- [Result] Ogasawara S, Mihara Y, Kondo R, Kusano H, Akiba J, Yano H. Antiproliferative Effect of Lenvatinib on Human Liver Cancer Cell Lines In Vitro and In Vivo. Anticancer Res. 2019 Nov;39(11):5973-5982. doi: 10.21873/anticanres.13802. PMID 31704822
- [Result] Ikeda K, Kudo M, Kawazoe S, Osaki Y, Ikeda M, Okusaka T, Tamai T, Suzuki T, Hisai T, Hayato S, Okita K, Kumada H. Phase 2 study of lenvatinib in patients with advanced hepatocellular carcinoma. J Gastroenterol. 2017 Apr;52(4):512-519. doi: 10.1007/s00535-016-1263-4. Epub 2016 Oct 4. PMID 27704266
- [Result] Alsina A, Kudo M, Vogel A, Cheng AL, Tak WY, Ryoo BY, Evans TRJ, Lopez Lopez C, Daniele B, Misir S, Ren M, Izumi N, Qin S, Finn RS. Effects of Subsequent Systemic Anticancer Medication Following First-Line Lenvatinib: A Post Hoc Responder Analysis from the Phase 3 REFLECT Study in Unresectable Hepatocellular Carcinoma. Liver Cancer. 2020 Jan;9(1):93-104. doi: 10.1159/000504624. Epub 2019 Dec 16. PMID 32071913
- [Result] Zhang BH, Cai YS, Jiang L, Yang JY. Donafenib as a first-line monotherapy for advanced hepatocellular carcinoma. Hepatobiliary Surg Nutr. 2021 Oct;10(5):737-740. doi: 10.21037/hbsn-21-304. No abstract available. PMID 34760990
- [Result] Qin S, Bi F, Gu S, Bai Y, Chen Z, Wang Z, Ying J, Lu Y, Meng Z, Pan H, Yang P, Zhang H, Chen X, Xu A, Cui C, Zhu B, Wu J, Xin X, Wang J, Shan J, Chen J, Zheng Z, Xu L, Wen X, You Z, Ren Z, Liu X, Qiu M, Wu L, Chen F. Donafenib Versus Sorafenib in First-Line Treatment of Unresectable or Metastatic Hepatocellular Carcinoma: A Randomized, Open-Label, Parallel-Controlled Phase II-III Trial. J Clin Oncol. 2021 Sep 20;39(27):3002-3011. doi: 10.1200/JCO.21.00163. Epub 2021 Jun 29. PMID 34185551
- [Derived] Zhou J, Tan Z, Sun B, Leng Y, Liu S. Application of indocyanine green fluorescence imaging in hepatobiliary surgery. Int J Surg. 2024 Dec 1;110(12):7948-7961. doi: 10.1097/JS9.0000000000001802. PMID 38884267